CLINICAL TRIAL: NCT05749016
Title: Neoadjuvant Inetetamab Combined With Pertuzumab and Paclitaxel/Carboplatin for Locally Advanced HER2-Positive Breast Cancer: a Prospective, Single-arm, Multi-center Phase II Study
Brief Title: Neoadjuvant Inetetamab Combined With Pertuzumab and Paclitaxel/Carboplatin for Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPNCb-01
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Locally Advanced Breast Cancer; Chemotherapy Effect
Keywords: Locally Advanced Breast Cancer; Neoadjuvant Chemotherapy
MeSH Terms: interventions — pertuzumab; Paclitaxel; Carboplatin; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The phase II trial included patients with histologically confirmed stage IIA to IIIC and HER2-positive primary invasive breast cancer from November 2021 to July 2023. Eligible patients received inetetamab with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen every three weeks for a maximum of 6 cycles, followed by surgery. The primary endpoint was pathologic complete response (pCR; ypT0 ypN0) rate. Key secondary endpoints included near pCR (npCR) (residual breast disease <1cm), objective response rate (ORR) and safety.
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study group (Experimental): Eligible patients received inetetamab with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen every three weeks for a maximum of 6 cycles, followed by surgery.
  Interventions: Drug: inetetamab with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen

INTERVENTIONS:
Drug: inetetamab with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen — Inetetamab (Cipterbin) is a newly marketed anti-HER2 monoclonal antibody with amino acid modified Fc region and enhanced antibody-dependent cellular cytotoxicity (ADCC) effect. There was no robust evidence evaluating the combination of inetetamab with pertuzumab and neoadjuvant chemotherapy (paclitaxel + carboplatin) in the neoadjuvant setting. This study aimed to evaluate the efficacy and safety of inetetamab + pertuzumab+paclitaxel + carboplatin (TCbIP) as a neoadjuvant chemotherapy regimen in the treatment of patients with locally advanced HER2-positive breast cancer.
  Other Names: Cipterbin with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen

SUMMARY:
Inetetamab (Cipterbin) is a newly marketed anti-HER2 monoclonal antibody with amino acid modified Fc region and enhanced antibody-dependent cellular cytotoxicity (ADCC) effect. There was no robust evidence evaluating the combination of inetetamab with pertuzumab and neoadjuvant chemotherapy (paclitaxel + carboplatin) in the neoadjuvant setting. This study aimed to evaluate the efficacy and safety of inetetamab + pertuzumab+paclitaxel + carboplatin (TCbIP) as a neoadjuvant chemotherapy regimen in the treatment of patients with locally advanced HER2-positive breast cancer.

DETAILED DESCRIPTION:
Inetetamab (Cipterbin) is a newly marketed anti-HER2 monoclonal antibody with amino acid modified Fc region and enhanced antibody-dependent cellular cytotoxicity (ADCC) effect. There was no robust evidence evaluating the combination of inetetamab with pertuzumab and neoadjuvant chemotherapy (paclitaxel + carboplatin) in the neoadjuvant setting. This study aimed to evaluate the efficacy and safety of inetetamab + pertuzumab+paclitaxel + carboplatin (TCbIP) as a neoadjuvant chemotherapy regimen in the treatment of patients with locally advanced HER2-positive breast cancer.

The phase II trial included female patients with histologically confirmed stage IIA to IIIC and HER2-positive primary invasive breast cancer. Eligible patients received inetetamab with pertuzumab and paclitaxel/carboplatin (TCbIP) regimen every three weeks for a maximum of 6 cycles, followed by surgery. The primary endpoint was pathologic complete response (pCR; ypT0 ypN0) rate. Key secondary endpoints included near pCR (npCR) (residual breast disease <1cm), objective response rate (ORR) and safety. Efficacy was analyzed in the intention-to-treat (ITT) and per-protocol (PP) populations. The ITT population included patients who received at least 2 cycles of the study drug but excluded those who were lost to follow-up without surgery and those who received other targeted therapy. The PP population was a subgroup of patients who met all the trial criteria, were compliant with the protocol, and did not violate any major protocols. Safety was analyzed in the safety population, which included all patients who received at least one dose of the study drug and had available safety data. Fisher's exact test was used for the comparisons between patients with pCR and those with non-pCR.

ELIGIBILITY:
Inclusion Criteria:

* Age of minimum of 18 years to a maximum of 70 years; males or females
* diagnosed as invasive breast carcinoma by preoperative needle core biopsy; patients with clinical stage of T1c to T4, N0-3, and M0, as defined by the American Joint Committee on Cancer AJCC Staging Manual, 8th Edition staging criteria
* HER2-positive: an immunohistochemistry (IHC) score of 3+ or IHC 2+ and in situ hybridization ISH+/fluorescence in situ hybridization FISH+.
* Left ventricular ejection fraction (LVEF) ≥50%；
* Eastern Cooperative Oncology Group (ECOG) performance score was 0/1；
* In the absence of blood transfusion or pharmacological treatment (granulocyte colony-stimulating factor/erythropoietin (EPO)/interleukin-11, etc.) within 14 days prior to the first treatment, and organ function must meet the following requirements: absolute neutrophil count (ANC) ≥ 1.5×109/L; platelets (PLT) ≥ 100×109/L; hemoglobin (Hb) ≥ 90g/L. Blood biochemistry: total bilirubin (TBIL) ≤1.5×ULN; ALT and AST ≤1.5×ULN; BUN and Cr ≤1.5×ULN; creatinine clearance ≥50mL/min (Cockcroft-Gault formula); total bilirubin (TBIL) ≤1.5×ULN; ALT and AST ≤1.5×ULN; BUN and Cr ≤1.5×ULN; creatinine clearance ≥50mL/min (Cockcroft-Gault formula);
* Volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

* had a previous history of invasive breast cancer;
* Bilateral breast cancer, inflammatory breast cancer (eg, erythema and/or skin involvement, and/or pathological findings of neoplastic cells in dermal lymphatic vessels);
* Previous excisional and/or excisional biopsy of primary tumor and/or axillary lymph nodes;
* Previous systemic therapy for breast cancer；
* History of previous life-threatening hypersensitivity reactions, or known hypersensitivity to any component of the study drug；
* Participated in clinical trials of other drugs or medical devices within 4 weeks before the first medication, and received treatment with experimental drugs or devices；
* Patients who have undergone major surgery within 28 days before the first dose, or plan to have major surgery during the study period；
* Other malignancies within the past 5 years (except cervical cancer in situ, non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ)；
* Active hepatitis, active tuberculosis or other serious infectious diseases, etc., including but not limited to: active hepatitis C virus (HCV) infection (except for HCV antibody positive but RNA negative), or active hepatitis B virus (HBV) infection (hepatitis B Surface antigen positive and HBV-DNA copy number >2000 IU/mL) or bacteremia, severe infectious pneumonia and other serious infections requiring systemic treatment
* History of immunodeficiency or other autoimmune diseases, including but not limited to human immunodeficiency virus (HIV) infection (HIV antibody positive), systemic lupus erythematosus, rheumatoid arthritis, or history of organ transplantation；
* Those with the following history of cardiovascular and cerebrovascular diseases, including: (1) unstable angina; (2) arrhythmia requiring drug treatment or clinically significant; (3) myocardial infarction within 6 months; (4) cardiac arrhythmia Failure, second-degree and above atrioventricular block; (5) cerebral infarction (except lacunar infarction), cerebral hemorrhage and other diseases within 6 months；
* Patients with poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg under regular drug control), or a history of hypertensive crisis or hypertensive encephalopathy；
* Pregnant and breastfeeding female patients; women of childbearing age who have a positive pregnancy test during the screening period; patients who are unwilling to take effective contraceptive measures during the entire test period and within 6 months after the end of the medication；
* Other conditions that the investigator considers inappropriate to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) rate | up to 6 months
  Proportion of patients with no residual invasive tumor cells on pathological examination of primary breast lesions and axillary lymph node surgical specimens of all patients

SECONDARY OUTCOMES:
near pathologic complete response | up to 6 months
  Proportion of patients with residual breast disease <1cm on pathological examination of primary breast lesions and axillary lymph node surgical specimens of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Binghe Xu, Dr., Study Director — National Cancer Center/National Clinical Research Center for Cancer
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Individual anonymized participant data will not be shared.

REFERENCES:
- [Derived] Jiang M, Chai Y, Liu J, He M, Wang Y, Yang X, Xing Z, Zhang M, Zhou S, Ma F, Wang J, Yuan P, Xu B, Li Q. Neoadjuvant inetetamab and pertuzumab with taxanes and carboplatin (TCbIP) In locally advanced HER2-positive breast cancer: a prospective cohort study with propensity-matched analysis. BMC Cancer. 2024 Jul 22;24(1):877. doi: 10.1186/s12885-024-12654-3. PMID 39039516